CLINICAL TRIAL: NCT03574376
Title: Protocol for a Single Center Randomized Controlled Trial of Liposomal Bupivacaine Intercostal Nerve Blockade Versus Continuous Thoracic Epidural for Regional Analgesia in Patients With Multiple Rib Fractures
Brief Title: Liposomal Bupivacaine Intercostal Nerve Block vs Thoracic Epidural for Regional Analgesia in Multiple Rib Fractures
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chadrick Evans (Other)
Collaborators: University of Illinois College of Medicine at Peoria (Other); OSF Healthcare System (Other)
Responsible Party: Sponsor-Investigator, Chadrick Evans, Director of Surgical ICU and Trauma, OSF Healthcare System
Organization: OSF Healthcare System (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1146837-2
Record Dates: First submitted 2018-06-01; First posted 2018-07-02 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Trauma; Trauma Injury; Pain, Acute
Keywords: Rib trauma, intercostal nerve block, liposomal bupivacaine
MeSH Terms: conditions — Wounds and Injuries; Accidental Injuries; Acute Pain | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: This is a two arm, randomized trial. Patients suffering multiple traumatic rib fractures will be offered CEA or LBINB. As the current standard of care, CEA will serve as the control, and outcomes measured in patients receiving LBINB will be statistically evaluated relative to the CEA control group.
  All patients will receive standardized NSAID and opioid analgesia protocol for break through pain, as well as standardized routines for pulmonary hygiene and physiotherapy.
Masking Description: No participants are blinded to treatment arms. Patients and investigators are aware of which patients are assigned to each treatment group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Bupivacaine Liposome Injection [Exparel] (Active Comparator): Patients will receive a nerve block with a medication called liposomal bupivacaine, also called Exparel. Once assigned, a University of Illinois surgeon, or resident surgeon, will administer the nerve block. The nerve block is expected to provide pain relief from 72 to 96 hours. During this time, patients may request oral or intravenous pain medication for breakthrough pain. Patients will remain in the hospital until discharged by the attending physician.
  Interventions: Drug: Bupivacaine Liposome Injection
- Epidural 0.125% bupivicaine (Active Comparator): Patients will receive pain relief through a 0.125% bupivacaine epidural in the upper back by an assigned anesthesiologist. This epidural will remain in place for an uncertain amount of time. The decision to remove the epidural will be determined by the physicians and will be based on level of pain and injury.
  However, pain data will only be recorded by the research team for no longer than 96 hours after the epidural is placed. Patients are able to request intravenous and oral pain medications for breakthrough pain. After the epidural is removed, they will remain in the hospital until discharged by the attending physician.
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine Liposome Injection — Under ultrasound guidance, corresponding ribs will be identified. 3-5 ml of a 1.3% (13.3 mg/mL) of liposomal bupivacaine will be drawn into a syringe with a 1.5-in, 22-gauge needle. The needle will then be advanced 20° cephalad to the skin 3-4 cm lateral to midline at the level of each fractured rib, and 1-2 ribs levels above and below injury. The needle will be advanced 3 mm below the inferior margin of the rib, placing the tip in the space containing the neurovascular bundle. Following negative aspiration for blood or air, 3-5 mL of local anesthetic will be infused and the needle withdrawn. No more than 266 mg, or 20 ml, of the 1.3% (13.3 mg/mL) liposomal bupivacaine solution will be injected
  Other Names: Exparel
  Arms: Bupivacaine Liposome Injection [Exparel]
Drug: Bupivacaine — The anesthesia department will manage CEA. If possible, the patient will be in the sitting position. The skin will be prepped with chlorhexidine and sterilely draped. 3 mL of lidocaine 1% will be infiltrated the closest interspace to the rib fractures between T4 -T12. A Touhy needle will be inserted, the epidural space identified by loss of resistance technique. An epidural catheter will then be inserted to a depth of 12cm. 3 mL of test solution with lidocaine 1.5% with epinephrine, 1:200,000 will be injected with continuous EKG and SpO2 monitoring. Delivery of a 0.125% bupivacaine solution be continuously infused and titrated based on the patient's clinical status
  Other Names: bupivacaine Hcl
  Arms: Epidural 0.125% bupivicaine

SUMMARY:
Management of traumatic rib fractures continues to be a challenge for trauma surgeons. Currently, many analgesic options are available to patients suffering from rib fractures. Formulations currently used for conventional intercostal nerve blocks (CINB) are relatively safe, do not require additional equipment or specialized anesthesia personnel, do not require catheter repositioning, and provide improved analgesia immediately over the aforementioned systemic therapies. A goal of these authors to introduce an additional safe option for extended local analgesia in the setting of multiple rib fractures given the inconclusive evidence supporting or refuting the current standard of care

DETAILED DESCRIPTION:
The objective of this study is to quantify and draw inferences on the efficacy of a multiple level liposomal bupivacaine intercostal nerve blockade (LBINB) in patients with multiple traumatic rib fractures.

The primary objective is to assess the quality and duration of analgesia based on numeric grading pain scale, improvement in pulmonary function parameters, reduction pulmonary complications, and duration of hospitalization in patients receiving LBINBs relative to those receiving the current standard of care, CEA, in patients recovering from multiple traumatic rib fractures.

The secondary objective of this study is to assess cost and rate of complications associated with LBINB relative to CEA.

This is a two arm, randomized trial. Patients suffering multiple traumatic rib fractures will be offered CEA or LBINB. As the current standard of care, CEA will serve as the control, and outcomes measured in patients receiving LBINB will be statistically evaluated relative to the CEA control group.

All patients will receive standardized NSAID and opioid analgesia protocol for break through pain, as well as standardized routines for pulmonary hygiene and physiotherapy.

Indications for CEA and LBINB in this study include patients suffering from traumatic thoracic injury with greater than or equal to 3 fractured ribs

ELIGIBILITY:
Inclusion Criteria:

* All patients 18 years of age or older suffering 3 or more rib fractures treated by University of Illinois College of Medicine at Peoria (UICOMP) attending or resident physicians at OSF St. Francis Medical Center (OSFMC) are potentially eligible for enrollment in the trial.

Exclusion Criteria:

* Patients with any of the following will not be eligible since they are contraindications to CEA, LBINB, or both:

  1. Intracranial hemorrhage
  2. Fever >101 degrees Fahrenheit for ≥ 1 hour(s)
  3. Rash at site of catheter insertion or administration of nerve block
  4. Hemodynamic instability
  5. Spinal cord injury
  6. Vertebral fractures
  7. Allergy to bupivacaine
  8. Systemic therapeutic anticoagulation required for duration of hospital admission 20
  9. Altered mental status without medical decision maker to provide consent
  10. Patients without the capacity to consent or the lack of a medical decision maker to consent
  11. Patients that are pregnant
  12. Legally confined patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Estimated)
Dates: Start 2018-08-29 (Actual); Primary Completion 2020-08-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in pain relief | 96 hours
  Quality of analgesia provided measured by numeric grading pain scale assessment every 24 hours over a 96-hour period. Pain will be rated using the Numerical Rating Scale, ranging from 0-10. Zero represents "no pain"; worsening pain signified by increasing reported numbers with 10 being the upper limit and the "worst pain possible". Only the numbers can be answers, meaning that there are only 11 possible answers on the 0-10 scale.

SECONDARY OUTCOMES:
Quantity of pain medication | 96 hours
  Amount of breakthrough analgesia required in morphine equivalents
Length of pain medication | every 24hours for 96hours
  Duration of analgesia provided measured by numeric grading pain scale assessment every 24hours. Quality of analgesia provided measured by numeric grading pain scale assessment every 24 hours over a 96-hour period. Pain will be rated using the Numerical Rating Scale, ranging from 0-10. Zero represents "no pain"; worsening pain signified by increasing reported numbers with 10 being the upper limit and the "worst pain possible". Only the numbers can be answers, meaning that there are only 11 possible answers on the 0-10 scale.
Pulmonary function | 96 hours
  Pulmonary function measured by incentive spirometry
Supplemental oxygen | 96 hours
  Supplemental oxygen requirements
Oxygen saturation | 96 hours
  Oxygen saturation levels
Pulmonary complications | 96 hours
  Development of pulmonary complications: atelectasis, pneumonia, respiratory failure
Ventilator | 96 hours
  Ventilator days
Overall length of stay | 96 hours
  Length of stay
ICU stay | 96 hours
  Duration of ICU days
Costs | 96 hours
  Costs associated with administration of epidural vs exparel
Overall complication rate | 96 hours
  Overall rate of complications associated with epidural vs exparel

CONTACTS AND LOCATIONS:
Overall Officials: Chadrick R Evans, MD, Principal Investigator — OSF Healthcare System
Locations (1):
- Osf St Francis Medical Center, Peoria, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ahn Y, Gorlinger K, Alam HB, Eikermann M. Pain-associated respiratory failure in chest trauma. Anesthesiology. 2013 Mar;118(3):701-8. doi: 10.1097/ALN.0b013e318283996b. No abstract available. PMID 23403516
- [Result] Battle CE, Hutchings H, Evans PA. Risk factors that predict mortality in patients with blunt chest wall trauma: a systematic review and meta-analysis. Injury. 2012 Jan;43(1):8-17. doi: 10.1016/j.injury.2011.01.004. Epub 2011 Jan 22. PMID 21256488
- [Result] Horlocker TT, Wedel DJ, Rowlingson JC, Enneking FK. Executive summary: regional anesthesia in the patient receiving antithrombotic or thrombolytic therapy: American Society of Regional Anesthesia and Pain Medicine Evidence-Based Guidelines (Third Edition). Reg Anesth Pain Med. 2010 Jan-Feb;35(1):102-5. doi: 10.1097/AAP.0b013e3181c15dd0. No abstract available. PMID 20048659
- [Result] Galvagno SM Jr, Smith CE, Varon AJ, Hasenboehler EA, Sultan S, Shaefer G, To KB, Fox AD, Alley DE, Ditillo M, Joseph BA, Robinson BR, Haut ER. Pain management for blunt thoracic trauma: A joint practice management guideline from the Eastern Association for the Surgery of Trauma and Trauma Anesthesiology Society. J Trauma Acute Care Surg. 2016 Nov;81(5):936-951. doi: 10.1097/TA.0000000000001209. PMID 27533913
- [Result] Rice DC, Cata JP, Mena GE, Rodriguez-Restrepo A, Correa AM, Mehran RJ. Posterior Intercostal Nerve Block With Liposomal Bupivacaine: An Alternative to Thoracic Epidural Analgesia. Ann Thorac Surg. 2015 Jun;99(6):1953-60. doi: 10.1016/j.athoracsur.2015.02.074. Epub 2015 Apr 23. PMID 25912739
- [Result] Nosotti M, Rosso L, Tosi D, Palleschi A, Mendogni P, Righi I, Marenghi C, Santambrogio L. Preventive analgesia in thoracic surgery: controlled, randomized, double-blinded study. Eur J Cardiothorac Surg. 2015 Sep;48(3):428-33; discussion 434. doi: 10.1093/ejcts/ezu467. Epub 2014 Dec 18. PMID 25527168
- [Result] Mohta M, Verma P, Saxena AK, Sethi AK, Tyagi A, Girotra G. Prospective, randomized comparison of continuous thoracic epidural and thoracic paravertebral infusion in patients with unilateral multiple fractured ribs--a pilot study. J Trauma. 2009 Apr;66(4):1096-101. doi: 10.1097/TA.0b013e318166d76d. PMID 19359920
- [Result] Khalil KG, Boutrous ML, Irani AD, Miller CC 3rd, Pawelek TR, Estrera AL, Safi HJ. Operative Intercostal Nerve Blocks With Long-Acting Bupivacaine Liposome for Pain Control After Thoracotomy. Ann Thorac Surg. 2015 Dec;100(6):2013-8. doi: 10.1016/j.athoracsur.2015.08.017. Epub 2015 Oct 24. PMID 26507422
- [Result] Karmakar MK, Critchley LA, Ho AM, Gin T, Lee TW, Yim AP. Continuous thoracic paravertebral infusion of bupivacaine for pain management in patients with multiple fractured ribs. Chest. 2003 Feb;123(2):424-31. doi: 10.1378/chest.123.2.424. PMID 12576361
- [Result] Battle CE, Hutchings H, James K, Evans PA. The risk factors for the development of complications during the recovery phase following blunt chest wall trauma: a retrospective study. Injury. 2013 Sep;44(9):1171-6. doi: 10.1016/j.injury.2012.05.019. Epub 2012 Jun 12. PMID 22695321
- [Result] Brasel KJ, Guse CE, Layde P, Weigelt JA. Rib fractures: relationship with pneumonia and mortality. Crit Care Med. 2006 Jun;34(6):1642-6. doi: 10.1097/01.CCM.0000217926.40975.4B. PMID 16625122
- [Result] Britt T, Sturm R, Ricardi R, Labond V. Comparative evaluation of continuous intercostal nerve block or epidural analgesia on the rate of respiratory complications, intensive care unit, and hospital stay following traumatic rib fractures: a retrospective review. Local Reg Anesth. 2015 Oct 27;8:79-84. doi: 10.2147/LRA.S80498. eCollection 2015. PMID 26604819
- [Result] Byun JH, Kim HY. Factors affecting pneumonia occurring to patients with multiple rib fractures. Korean J Thorac Cardiovasc Surg. 2013 Apr;46(2):130-4. doi: 10.5090/kjtcs.2013.46.2.130. Epub 2013 Apr 9. PMID 23614099
- [Result] Carrier FM, Turgeon AF, Nicole PC, Trepanier CA, Fergusson DA, Thauvette D, Lessard MR. Effect of epidural analgesia in patients with traumatic rib fractures: a systematic review and meta-analysis of randomized controlled trials. Can J Anaesth. 2009 Mar;56(3):230-42. doi: 10.1007/s12630-009-9052-7. Epub 2009 Feb 11. PMID 19247744
- [Result] Dehghan N, de Mestral C, McKee MD, Schemitsch EH, Nathens A. Flail chest injuries: a review of outcomes and treatment practices from the National Trauma Data Bank. J Trauma Acute Care Surg. 2014 Feb;76(2):462-8. doi: 10.1097/TA.0000000000000086. PMID 24458051
- [Result] Duch P, Moller MH. Epidural analgesia in patients with traumatic rib fractures: a systematic review of randomised controlled trials. Acta Anaesthesiol Scand. 2015 Jul;59(6):698-709. doi: 10.1111/aas.12475. Epub 2015 Feb 13. PMID 25683770
- [Result] Ho AM, Karmakar MK, Critchley LA. Acute pain management of patients with multiple fractured ribs: a focus on regional techniques. Curr Opin Crit Care. 2011 Aug;17(4):323-7. doi: 10.1097/MCC.0b013e328348bf6f. PMID 21716105
- [Result] Hwang EG, Lee Y. Effectiveness of intercostal nerve block for management of pain in rib fracture patients. J Exerc Rehabil. 2014 Aug 31;10(4):241-4. doi: 10.12965/jer.140137. eCollection 2014 Aug. PMID 25210700
- [Result] Ilfeld BM, Malhotra N, Furnish TJ, Donohue MC, Madison SJ. Liposomal bupivacaine as a single-injection peripheral nerve block: a dose-response study. Anesth Analg. 2013 Nov;117(5):1248-56. doi: 10.1213/ANE.0b013e31829cc6ae. PMID 24108252
- [Result] Ilfeld BM, Viscusi ER, Hadzic A, Minkowitz HS, Morren MD, Lookabaugh J, Joshi GP. Safety and Side Effect Profile of Liposome Bupivacaine (Exparel) in Peripheral Nerve Blocks. Reg Anesth Pain Med. 2015 Sep-Oct;40(5):572-82. doi: 10.1097/AAP.0000000000000283. PMID 26204387
- See also: Management of Antithrombotic Therapy for Neuraxial and Peripheral Nerve Procedures — https://depts.washington.edu/anticoag/home/content/neuraxial-guidelines

DOCUMENTS (2):
  • Informed Consent Form (2017-05-10): https://cdn.clinicaltrials.gov/large-docs/76/NCT03574376/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2017-06-05): https://cdn.clinicaltrials.gov/large-docs/76/NCT03574376/Prot_SAP_001.pdf